CLINICAL TRIAL: NCT02230787
Title: Effect of Emdogain on Wound Healing After Gingival Recession Coverage Using Connective Tissue Graft: A Pilot Study
Brief Title: Gingival Recession Coverage With and Without Emdogain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 186/13
Record Dates: First submitted 2014-08-12; First posted 2014-09-03 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Gingival Recession; Emdogain
Keywords: Pilot study; randomized clinical trial; periodontal disease; gingival recession; Emdogain; connective tissue; wound healing; inflammation
MeSH Terms: conditions — Gingival Recession; Periodontal Diseases; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Recession coverage without Emdogain (Active Comparator)
  Interventions: Device: Recession coverage without Emdogain
- Recession coverage with Emdogain (Experimental)
  Interventions: Device: Recession coverage with Emdogain

INTERVENTIONS:
Device: Recession coverage without Emdogain — In the control group subjects the recession coverage surgery will be performed without Emdogain.
  Arms: Recession coverage without Emdogain
Device: Recession coverage with Emdogain — In the test group subjects the recession coverage surgery will be performed with Emdogain.
  Arms: Recession coverage with Emdogain

SUMMARY:
Enamel matrix proteins have been shown to play a crucial role during tooth development and its supporting tissues. This is used in periodontal surgery where regeneration of lost tissues around the teeth is intended. Emdogain, a product of Straumann Institute contains these matrix proteins and has been successfully used in regenerative periodontal surgery for more than 16 years.

The treatment of gum recession is a common requirement, more and more patients are seeking treatment at the investigators' clinic due to aesthetic concern, root sensitivity and difficulties in performing adequate oral hygiene. The standard treatment comprises the transplantation of a piece of connective tissue from the palate to the denuded root surface. In many cases Emdogain is additionally applied to enhance healing. So far the effect of Emdogain on the early wound healing process after surgical root coverage has not been investigated.

The purpose of the investigators' study is to compare early wound healing parameters between treatment with and without Emdogain. For this study 40 patients undergoing root coverage surgery at the investigators' department will be included. Early wound healing features between the two groups will be described and compared. Furthermore, inflammatory markers typical for early healing will be evaluated together with patients'subjective postoperative comfort. Finally, outcomes 6 months after the treatment will be assessed. The investigators' hypothesis is that Emdogain treatment enhances wound healing and decreases post-operative complication rates.

DETAILED DESCRIPTION:
Background

Effect of Emdogain on wound healing after gingival recession coverage using connective tissue graft: a pilot study Emdogain Treatment Emdogain (Institute Straumann, Basel Switzerland) is an enamel matrix protein derivative with the vehicle propylene glycol alginate. Emdogain has been used for more than 16 years for regenerative periodontal treatment of intrabony, class II furcation and recession defects. Animal and human histological studies have provided evidence for periodontal regeneration (e.g. formation of root cementum, periodontal ligament and alveolar bone) following the application of Emdogain in conjunction with periodontal surgery. The use of Emdogain has been shown to significantly improve the clinical outcomes evidenced by probing depth reduction, and clinical attachment gain and is considered today as a routine procedure.

Background Therapy of buccal gingival recession is a common indication for treatment in order to improve plaque control thus preventing gingivitis and root caries but also to improve aesthetics and root sensitivity. The ultimate goal of a root coverage procedure is the complete coverage of the root surface and, in the same time, to obtain a similar appearance of the regenerated soft tissues to the surrounding intact tissues. The use of palatal connective tissue graft in conjunction with a coronally advanced flap (CAF) is a well established clinical procedure for the treatment of gingival recessions. Its use has been shown to result in predictable root coverage, higher increase in keratinized tissue and more stable long-term outcomes compared to the use of CAF and is considered today state of the art. Furthermore, recent data also appear to indicate that the combination of Emdogain and CTG may additionally improve the clinical outcomes. Therefore, the standard surgical procedure for the treatment of gingival recessions at the Department of Periodontology includes the use of connective tissue graft either with or without the use of Emdogain.

Interestingly, despite the fact that Emdogain is commonly used, no information on its effects upon early wound healing is available.

Hence, the aim of this study is to evaluate the effect of Emdogain on early wound healing, as assessed by means of clinical parameters and inflammatory markers following recession coverage surgery.

Study population and methodology Patient groups compared: in the treatment group, patients undergoing a recession coverage surgery will be treated with Emdogain whereas in the control group, patients will not receive Emdogain. A total of 40 patients, 20 in each group will be included.

Preoperative inflammatory markers will be assessed at the preoperative examination and two days after surgery by dipping paper points into the crevicular fluid. Furthermore the investigators will assess whether remnants of Emdogain are still traceable two days after surgery. Wound healing after root coverage procedure is assessed using the "early wound healing index (EHI)" defined by Wachtel et al. According to Wachtel et al., wound healing is quantified and graded into 5 stages.

Additionally, the post-operative healing process will be judged by a patient questionnaire. Finally root coverage is measured as the distance from the CEJ (Cemento Enamel Junction) to the Margo Gingivae in mm.

Objective

1. To investigate the benefit of intraoperative use of Emdogain on early wound healing during the first two weeks after gingival recession coverage. Early wound healing parameters will be assessed at both the site of explantation of the tissue graft as well as at the site of implantation.
2. To investigate the effect of Emdogain on inflammatory markers in crevicular fluid and whether Emdogain is traceable after two days after application.
3. To investigate its influence on post-operative pain and interference with daily activities during the first two weeks (patient's questionnaire).
4. The post-operative result will also be assessed after 6 months.

Methods

The present prospective study will include a total of 40 patients, 20 patients in each of the 2 groups (Emdogain group and control group). All procedures will be elective procedures. After oral and written informed consent, the study will comprise the collection of crevicular fluid sampling and clinical data as well as the filling of a patient questionnaire. The study will be conducted as randomized prospective study. In the treatment group the procedure will be performed with Emdogain, in the control group, root coverage will be performed without, respectively. All procedures will be performed by one experienced operator. Patients will all be treated with the standard surgical procedure of the University of Bern. In the patient group with Emdogain, tissue graft and explantation site will be covered with Emdogain, in the patient group without Emdogain, no Emdogain will be used. After inclusion of the patients, the study duration will last 6 months for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Gingival recession Miller class I and II
* Written informed consent

Exclusion Criteria

* Patients with a history of a chronic infectious or inflammatory diseases (i.e. rheumatoid arthritis, systemic lupus erythematodes, Crohn's disease, or HIV-, HCV-infection etc.
* Patients with any clinical signs of an acute infection
* Patients with renal failure (GFR < 30ml/min)
* Smoking > 5 cigarettes per day
* Patients < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-04-22 (Actual); Study Completion 2017-02-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in wound healing | 2, 7 and 14 days after surgery
  Progress in wound healing assessed by the "early wound healing index (EHI)" previously defined by Wachtel et al.

SECONDARY OUTCOMES:
Levels of post-procedural inflammatory markers | 2 and 7 days after surgery
  Including IL- 8, IL-10, IL-1beta, MMP-8 and TGF beta-1, traceability of Emdogain in the operation field
Improvement of patients' post-operative comfort | 2 days to 2 weeks after surgery
  Assessed by patient questionnaire
Root coverage | 6 months after surgery
  Measured in mm

CONTACTS AND LOCATIONS:
Overall Officials: Anton Sculean, Prof. Dr. med. dent., Principal Investigator — Department of Periodontology, University of Bern
Locations (1):
- Department of Periodontology, University of Bern, Bern, Switzerland

REFERENCES:
- [Background] Grandin HM, Gemperli AC, Dard M. Enamel matrix derivative: a review of cellular effects in vitro and a model of molecular arrangement and functioning. Tissue Eng Part B Rev. 2012 Jun;18(3):181-202. doi: 10.1089/ten.TEB.2011.0365. Epub 2011 Dec 28. PMID 22070552
- [Background] Spahr A, Haegewald S, Tsoulfidou F, Rompola E, Heijl L, Bernimoulin JP, Ring C, Sander S, Haller B. Coverage of Miller class I and II recession defects using enamel matrix proteins versus coronally advanced flap technique: a 2-year report. J Periodontol. 2005 Nov;76(11):1871-80. doi: 10.1902/jop.2005.76.11.1871. PMID 16274306
- [Background] Wachtel H, Schenk G, Bohm S, Weng D, Zuhr O, Hurzeler MB. Microsurgical access flap and enamel matrix derivative for the treatment of periodontal intrabony defects: a controlled clinical study. J Clin Periodontol. 2003 Jun;30(6):496-504. doi: 10.1034/j.1600-051x.2003.00013.x. PMID 12795787
- [Background] Cairo F, Pagliaro U, Nieri M. Treatment of gingival recession with coronally advanced flap procedures: a systematic review. J Clin Periodontol. 2008 Sep;35(8 Suppl):136-62. doi: 10.1111/j.1600-051X.2008.01267.x. PMID 18724847
- [Result] Henriques PS, Pelegrine AA, Nogueira AA, Borghi MM. Application of subepithelial connective tissue graft with or without enamel matrix derivative for root coverage: a split-mouth randomized study. J Oral Sci. 2010 Sep;52(3):463-71. doi: 10.2334/josnusd.52.463. PMID 20881341
- [Result] Cueva MA, Boltchi FE, Hallmon WW, Nunn ME, Rivera-Hidalgo F, Rees T. A comparative study of coronally advanced flaps with and without the addition of enamel matrix derivative in the treatment of marginal tissue recession. J Periodontol. 2004 Jul;75(7):949-56. doi: 10.1902/jop.2004.75.7.949. PMID 15341352
- [Result] Aroca S, Molnar B, Windisch P, Gera I, Salvi GE, Nikolidakis D, Sculean A. Treatment of multiple adjacent Miller class I and II gingival recessions with a Modified Coronally Advanced Tunnel (MCAT) technique and a collagen matrix or palatal connective tissue graft: a randomized, controlled clinical trial. J Clin Periodontol. 2013 Jul;40(7):713-20. doi: 10.1111/jcpe.12112. Epub 2013 Apr 30. PMID 23627374
- [Result] Rasperini G, Roccuzzo M, Francetti L, Acunzo R, Consonni D, Silvestri M. Subepithelial connective tissue graft for treatment of gingival recessions with and without enamel matrix derivative: a multicenter, randomized controlled clinical trial. Int J Periodontics Restorative Dent. 2011 Apr;31(2):133-9. PMID 21491012